CLINICAL TRIAL: NCT01662128
Title: Randomized Controlled Trials of Efficacy and Safety With Xeloda as Sequential Adjuvant Therapy After Chemotherapy of Anthracycline and/or Taxane in Breast Cancer of Triple Negative or HER-2 Positive or Axillary Lymph Node Metastasis ≥4
Brief Title: Efficacy and Safety Of Xeloda as Sequential Adjuvant Therapy After Chemotherapy in Breast Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University (Other)
Responsible Party: Principal Investigator, Zhang jin, Professor, Tianjin Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: xeloda
Record Dates: First submitted 2012-08-02; First posted 2012-08-10 (Estimated); Last update posted 2012-08-10 (Estimated); Status verified 2012-08

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Xeloda (Experimental): Xeloda
  Interventions: Drug: Xeloda

INTERVENTIONS:
Drug: Xeloda — Xeloda as Adjuvant Therapy

SUMMARY:
Select 600 cases of women with breast cancer of triple negative or Her-2 positive or with more than 4 axillary lymph node metastasis. All the patients were accepted the chemotherapy of Anthracycline and/or Taxane. Divide them into two groups randomly. Then the experimental group will be treated with Xeloda(1000mg/m2,orally,2 times/day) for six cycles (21 days/cycle,each taking two weeks suspending for one week) as Sequential Adjuvant Therapy. And the control group will not receive any adjuvant therapy.Finally the investigators will assess the 5-year disease-free survival, 5 years and 10-year overall survival and safety of using medications.

DETAILED DESCRIPTION:
The investigators will select 600 cases of women with breast cancer of triple negative or Her-2 positive or with more than 4 axillary lymph node metastasis. All the patients were accepted the chemotherapy of Anthracycline and/or Taxane. Divide them into two groups randomly. Then the experimental group will be treated with Xeloda(1000mg/m2,orally,2 times/day) for six cycles (21 days/cycle,each taking two weeks suspending for one week) as Sequential Adjuvant Therapy. And the control group will not receive any adjuvant therapy.Finally the investigators will assess the 5-year disease-free survival, 5 years and 10-year overall survival and safety of using medications.

ELIGIBILITY:
Inclusion Criteria:

1. Karnofsky ≥ 70
2. Provision of informed consent
3. Pathological confirmation of breast cancer and exclusion of other metastases.
4. Pathological confirmation of triple negative or Her-2 positive or with more than 4 axillary lymph node metastasis
5. The patients have finished the chemotherapy of Anthracycline and/or Taxane.And it's no more than 28 days from accepting the last chemotherapy.
6. Laboratory criteria:

PLT ≥ 100*109/L WBC ≥ 4000/mm3 HGB ≥ 10g/dl GOT,GPT,ALP ≤ 2*ULN TBIL,DBIL,CCr ≤ 1.5*ULN

Exclusion Criteria:

1. Pregnant or lactation woman
2. Bilateral breast cancer, inflammatory breast cancer or carcinoma in situ
3. Accepted neoadjuvant treatment including chemotherapy, radiotherapy and endocrine therapy
4. History of organ transplantation
5. With mental disease
6. With severe infection or active gastrointestinal ulcers
7. With severe liver disease (such as cirrhosis), kidney disease, respiratory disease or diabetes
8. Disease-free period of other malignant tumor is less than 5 years(except cured basal cell skin cancer and cervical carcinoma in situ)
9. With heart disease
10. Experimental drug allergy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2012-06; Primary Completion 2014-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Adverse reactions | 6 months
  The occurrence of adverse reactions and the number of cases

SECONDARY OUTCOMES:
Disease-free survival | 5 years
  Disease-free survival of 5 years

OTHER OUTCOMES:
Overall survival,recurrence or death | 10 years
  Overall survival,recurrence or death of 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Jin Zhang, Professor, Study Chair — Tianjin Cancer Hospital
Locations (1):
- Tianjin Cancer Hospital, Tianjin, Tianjin Municipality, China